CLINICAL TRIAL: NCT03108729
Title: An Open-label Eslicarbazepine Acetate Long-term Safety and Tolerability Study in Children and Adolescents (4 - 17 Years)
Brief Title: A Pediatric Drug Study to Determine the Long-term Safety and Tolerability in Children and Adolescents (4-17 Years in Age) Taking the Drug
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not withdrawn for safety reasons. The sponsor received approval for the treatment of partial-onset seizures in patients 4 years of age and older
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP-093-364
Record Dates: First submitted 2017-03-27; First posted 2017-04-11 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Epilepsy
Keywords: epilepsy; Partial-onset seizures; Focal epilepsy; Focal seizures; Partial onset seizures; Pediatric; Partial seizures
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures | interventions — eslicarbazepine acetate

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- eslicarbazepine acetate (Experimental): elicarbazepine acetate, once daily flexible dosing
  Interventions: Drug: Eslicarbazepine acetate

INTERVENTIONS:
Drug: Eslicarbazepine acetate — Eslicarbazepine acetate tablets, taken once daily for 1 year. The daily maintenance dose will be within the range of 300 mg to 1600 mg ESL, and is determined by body weight, clinical response and tolerability.
  Other Names: Aptiom; ESL; SEP-0002093; BIA 2-093

SUMMARY:
A pediatric drug study to determine the long-term safety and tolerability in children and adolescents (4-17 years in age) taking the drug (elsicarbazepine acetate)

DETAILED DESCRIPTION:
This is a long-term, multicenter, open-label, safety, tolerability, and maintenance of effect study of flexible daily dosing with Eslicarbazepine acetate (ESL) in subjects 4 to 17 years of age with partial onset seizures (POS). The study is designed to enroll subjects to receive ESL as adjunctive treatment with the option to convert to ESL monotherapy after 6 months of ESL adjunctive treatment. Approximately 150 subjects will be enrolled to obtain approximately 75 subjects completing 1 year of treatment. At least 25% of subjects will be enrolled in each age group (4 - 6, 7 - 11, and 12 - 17 years of age). An attempt will be made to enroll no fewer than 30% of subjects in each gender. It is anticipated that approximately 50 subjects will convert to monotherapy during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 4 to < 18 y at enrollment, and weighs at least 11 kg at Screening and on the first day of ESL dosing.
2. The informed consent must be signed by the parent or legal guardian, and, when appropriate and/or required by state or local law, minor subjects must give written informed assent prior to participation in the study. All subjects in the United States (US) must have a parent or legal guardian, sign a Health Insurance Portability and Accountability Act (HIPAA) form.
3. Confirmed diagnosis of epilepsy with partial onset seizures as defined in the Classification of Seizures of the International League Against Epilepsy:

   1. Epilepsy with partial onset seizures with observable motor component, or complex partial seizures, with or without secondary generalization
   2. Documented EEG recording without generalized epileptiform abnormalities and with demonstrated focal abnormalities (done within 5 years prior to screening)
4. Documented magnetic resonance imaging (MRI) scan conducted within 5 years (older scans may be acceptable with consent of Medical Monitor) prior to screening, showing either normal results or static focal abnormalities.
5. Documented seizure frequency of at least 6 seizures per month prior to screening as reported by a caregiver and documented in subject's seizure history. Note: Retrospective reporting of seizure frequency does not require diary documentation.
6. Stable treatment with 1 to 3 AEDs (excluding carbamazepine and oxcarbazepine) for ≥ 2 weeks prior to screening and at least 4 weeks prior to the first ESL dose. Vagal nerve stimulation (if present) does not count as an AED.
7. Subject and/or caregiver are willing and able to complete a daily seizure diary for the duration of the study and comply with study procedures.
8. A female subject is eligible to enter and participate in the study if she is of:

   1. Non-childbearing potential because she is premenarchal (as assessed by physical examination) and < 7 y; or
   2. Non-childbearing potential because she is premenarchal (as assessed by physical examination), ≥ 7 y, and has a negative urine pregnancy test at screening; or
   3. Childbearing potential; has a negative serum pregnancy test at screening and agrees to satisfy one of the following requirements:

      • Complete abstinence from intercourse as a component of a habitually abstinent lifestyle; a minimum of 4 weeks prior to administration of the first dose of study drug, throughout the treatment period, and for a minimum of 8 weeks after completion or premature discontinuation from the study drug (abstinence must be part of an established abstinent lifestyle), and agrees to use a double-barrier method if she becomes sexually active; or

      • Established use of acceptable methods of contraception; a minimum of 4 weeks prior to administration of the first dose of study drug, throughout the treatment period, and for a minimum of 8 weeks after completion or premature discontinuation from the study drug. Acceptable methods of birth control are those with established failure rates of < 1%per year and include:
      * Double barrier birth control, which is limited to a condom plus spermicide or a condom plus diaphragm.
      * Intrauterine device (IUD). Note: Female subjects who are ≥ 7 y and premenarchal will not routinely undergo serum pregnancy tests and will only be administered a urine pregnancy test. A positive urine pregnancy test should be confirmed by a serum test in these subjects regardless of weight. Female subjects who are < 7 y will not undergo a serum or a urine pregnancy test.

   Note: ESL may interfere with the action of hormonal contraceptive and therefore hormonal contraceptives are not sufficient for this protocol.
9. Males must be willing to remain sexually abstinent (consistent with lifestyle) or use an effective method of birth control (eg, male using condom and female using diaphragm, contraceptive sponge, spermicide, contraceptive pill, or intrauterine device) from signing informed consent to at least 7 days after the last dose of study drug has been taken.
10. Stable environment with caregiver who can assist in completion of seizure diary and other study assessments, if needed.
11. Subject and/or caregiver must read and write and possess an educational level and degree of understanding of the local language at a level sufficient to complete study related assessments or communicate suitably with the Investigator and study coordinator. For subjects who do not meet this criterion, a caregiver must be able to meet this requirement on the subject's behalf.

Inclusion Criteria for Monotherapy Conversion Subjects (at or after Month 6)

1. Subject is < 18 years-old at time of taper/conversion.
2. Subject has a satisfactory response to ESL at ≥ 6months of treatment in present study (based on tolerability and reduction in seizures, as determined by the Investigator).
3. Subject is receiving 1 or 2 background AEDs (not including benzodiazepine or barbiturate).
4. Subject does not have history of status epilepticus in the previous 3 years.

Exclusion Criteria:

1. Subject has had prior exposure to or previously participated in a clinical study with ESL.
2. Subject has a history of allergic reaction to oxcarbazepine or carbamazepine, or a history of serious allergic reaction (Stevens Johnson syndrome, Drug Reaction with Eosinophilia and Systemic Symptoms [DRESS] or similar) to any AED, or a history of serious allergic reactions to other medications.
3. Subject has had an EEG showing generalized discharges.
4. Subject has had any of the following seizure types at any time: myoclonic, absence, or atonic.
5. Subject has Lennox-Gastaut Syndrome or other secondary generalized epilepsy (including inborn errors of metabolism), or Benign Rolandic Epilepsy.
6. Subject has a current diagnosis or a history of psychogenic seizures.
7. Subject has current seizures related to an acute medical illness.
8. Subject has purely subjective seizures.
9. Subject has had status epilepticus while taking any seizure medicine in the 3 years prior to screening.
10. Subject should not have had febrile illness ≤ 2 weeks prior to screening.
11. Subject is currently taking more than 3 AEDs or is taking carbamazepine or oxcarbazepine.
12. Subject is taking any protocol-prohibited medication within 4 weeks of first ESL dose.
13. Subject has any confounding factor such as pseudoseizures or syncope.
14. Subject has a known progressive structural CNS lesion(s) or progressive encephalopathy.
15. Subject (≥ 6 y) has an active suicidal plan or intent (in the Investigator's opinion) in the past 4 weeks prior to screening.
16. Subject has a history of suicide attempt in the last 2 years prior to screening.
17. Subject is at imminent risk of suicidal or homicidal action (in the Investigator's opinion).
18. Subjects who meet the Diagnostic and Statistical Manual of Mental Disorders, 5th edition text revision (DSM-V-TR) defined criteria for major depressive episode (MDE) within the last 6 months. Subjects with mild, chronic depression without recent hospitalization who are being maintained on a stable dose of a single antidepressant are acceptable.
19. Subject has a significant psychiatric disorder or history of recurrent episodes of severe depression requiring pharmacologic treatment or hospitalization within 2 years prior to screening.
20. Subject has a history of alcohol or substance abuse within 2 years prior to screening for study participation, or subjects currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medication in a manner, which, in the opinion of the Investigator, indicates abuse. Subjects who are regular users of medical marijuana are excluded; use during participation is prohibited.
21. Subject has a positive urine drug screen (UDS) at screening. Note: Subjects with a positive drug screen for amphetamines, opiates, or benzodiazepines, who have a prescribed medication for at least 4 weeks prior to screening, may be eligible to participate in the study upon approval from the Medical Monitor.
22. Subject has a major medical illness other than epilepsy that would prevent safe participation in this study, at the discretion of the Investigator, such as (but not limited to) chronic liver or kidney impairment.
23. Subject has a disorder or history of a condition that may interfere with drug absorption, distribution, metabolism, or excretion (eg, malabsorption, gastrointestinal surgery, clinically significant abnormality of the hepatic or renal system). Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Monitor should be consulted.

Subject has a history or presence of abnormal ECG, which in the Investigator's opinion is clinically significant or QTcB of ~ 450 msec per screening central over read ECG.

25. Subject is known to have tested seropositive for the human immunodeficiency virus (HIV).

26. Subject has a positive history for the hepatitis B surface antigen or hepatitis C antibody.

27. Subject has a history of hypothyroidism, hyperthyroidism, or has values for thyroid testing (free T3, free T4, thyroid stimulating hormone [TSH]) indicating the presence of significant thyroid dysfunction.

28. Subjects has the following abnormal laboratory tests (not limited to, but including the following): a. Aspartate aminotransferase (ALT)/alanine aminotransferase (AST) > 1.5 times the upper limit of normal (ULN) b. White blood cell (WBC) count of < 2500 cells/μL c. Platelet count of < 100 × 103 cells/μL

Note: Subjects with stable platelet counts over the last 3 months prior to screening in the range of 80 × 103 to 100 × 103 cells/μL are eligible to participate in the study.

d. Subjects have estimated creatinine clearance by modified Schwartz GFR of 77.8 mL/min/1.73m2.

e. Subject has a sodium level of < 130 mEq/L.

Note: If any laboratory exclusion criteria are outside the normal range, the necessity for a repeat test should be discussed with the Medical Monitor. If upon retesting the value remains outside the protocol-specified range, the significance of this value may be discussed with the Medical Monitor for enrollment consideration.

29. Subject has difficulty providing blood samples due to poor venous access or cannot safely provide a sufficient quantity of blood.

30. Subjects of Asian ancestry must not be carriers of HLA b*1502. Either: a) subjects/caregivers must give written informed consent for genotyping, and test negative, or b) subjects/caregivers must provide documentation of prior testing confirming non carrier status and documented in subject's medical history.

31. Subject is a female who is currently breastfeeding or intending to breastfeed during the study period, or within 3 months postpartum at the time of signing informed consent.

32. Subject has participated in any investigational study within 30 days prior to screening, as documented in subject's medical history.

33. Subject is unable to comply with study visit schedules or study procedures, except those that can be performed by a caregiver.

34. Subject is a Clinical or Investigational Site staff member or relative of a staff member.

35. Subject has experienced significant blood loss within 60 days or has donated plasma within 72 hours prior to Visit 1 or intends to donate blood or undergo elective surgery during the study or within 60 days following the study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs). | From the time the informed consent is signed to the end of the study, assessed up to 2 years
  Number of subjects with adverse events (AEs).
Percentage of subjects with adverse events (AEs). | From the time the informed consent is signed to the end of the study, assessed up to 2 years
  Percentage of subjects with adverse events (AEs).
Number of subjects with serious adverse events (SAEs). | From the time the informed consent is signed to the end of the study, assessed up to 2 years
  Number of subjects with serious adverse events (SAEs).
Percentage of subjects with serious adverse events (SAEs). | From the time the informed consent is signed to the end of the study, assessed up to 2 years
  Percentage of subjects with serious adverse events (SAEs).
Number of subjects with adverse events (AEs) leading to discontinuation. | From the time the informed consent is signed to the end of the study, assessed up to 2 years
  Number of subjects with adverse events (AEs) leading to discontinuation.
Percentage of subjects with adverse events (AEs) leading to discontinuation. | From the time the informed consent is signed to the end of the study, assessed up to 2 years
  Percentage of subjects with adverse events (AEs) leading to discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: CNS Mecdical Director, Study Director — Sunovion Pharmacetuicals Inc.
Locations (1):
- Child Neurology Specialists / Clinical Research Center of Nevada, LLC, Henderson, Nevada, United States